CLINICAL TRIAL: NCT02311023
Title: A Single Centre Open Six Months Study of Intermittent Fasting for the Treatment of People With Refractory Epilepsy.
Brief Title: Intermittent Fasting in Refractory Epilepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties recruiting
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Dr Alan Wah Cheong Yuen, Honorary Research Associate, University College London Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCLH 13/0389
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intermittent fasting (Experimental): Patients consume their normal diet for 5 days in the week. On 2 days they only consume 500 Cals if female and 600 Cals if male.
  Interventions: Other: Intermittent fasting

INTERVENTIONS:
Other: Intermittent fasting

SUMMARY:
This is an open trial of intermittent fasting in a group of patients with refractory seizures. Patients will continue on the diet for 6 months to assess the impact of the diet on seizure frequency.

DETAILED DESCRIPTION:
A proportion of people with epilepsy continue to have seizures despite all conventional treatment options. The classical ketogenic diet and its variants have been shown to help some of these people. However, these diets require significant medical and dietician supervision,and is frequently not well tolerated. There is a need to develop other diet therapy that is easier to administer and more acceptable to the patient. This trial undertaken in adult overweight UCLH outpatients examines the effect of an intermittent fasting diet on seizures. Subjects may consume their normal diet for 5 days a week. On 2 days in a week, they consume only 25% of their daily calorie requirement. Subjects will continue on the diet for 6 months. Intermittent fasting has been shown in animal studies to activate a number of signalling pathways which are thought to reduce seizure thresholds. Has intermittent fasting in humans might be expected to reduce seizures.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing at least 2 seizures per month
* .BMI of 25 or over

Exclusion Criteria:

* Current/previous eating disorder
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Daily total number of seizures | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- UCLH , The Epilepsy Society, Chalfont Saint Peters, Buckinghamshire, United Kingdom